CLINICAL TRIAL: NCT00962533
Title: A Two-year, Randomized, Controlled, Open-label, Virologic Response Adaptive Design, Multicenter Study to Optimize Antiviral Efficacy of Telbivudine in Adult Patients With HBeAg Positive Chronic Hepatitis B (EFFORT Study)
Brief Title: EFFicacy Optimization Research of Telbivudine Therapy
Acronym: EFFORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Major Science and Technology Special Project of China Eleventh Five-year (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH-01
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-03

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ROADMAP Group (Group I) (Experimental): Patients were to take telbivudine 600 mg orally daily from Baseline.At Week 24, patients in Group I were split into Group I-A or Group I-B based on their virologic load:
  * Group I-A: This group of patients was those with HBV DNA ≥300 copies/mL at Week 24 and adefovir was to be added at Week 28;
  * Group I-B: This group of patients was those with HBV DNA <300 copies/mL at Week 24. Telbivudine monotherapy was to be continued until there was a viral breakthrough (confirmed by two examinations with at least 1 month interval with compliance factor excluded) and then adefovir was to be added;
  The total treatment duration was 104 weeks.
  Interventions: Drug: telbivudine
- SOC (Standard of Care) Group (Group II) (Active Comparator): patients were to take telbivudine 600 mg monotherapy from Baseline until Week 104. If viral breakthrough (defined as HBV DNA 1 log10 above nadir) was confirmed (by two examinations with at least a 1 month interval with compliance factor excluded), adefovir 10 mg daily was to be added.
  Interventions: Drug: telbivudine

INTERVENTIONS:
Drug: telbivudine — telbivudine, 600mg, oral, daily
  Other Names: Sebivo®
  Arms: ROADMAP Group (Group I)
Drug: telbivudine — telbivudine, 600mg, oral, daily
  Other Names: Sebivo®
  Arms: SOC (Standard of Care) Group (Group II)

SUMMARY:
The purpose of this trial is to prove that the strategy of treatment adjustment at W24 according to virological response based on ROADMAP concept is better than standard of care strategy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, from 18 (inclusive) to 65 (inclusive) years of age
* HBsAg and HBeAg positive for over six months
* Patient is willing and able to comply with the study drug regimen and all other study requirements
* Patients must give written informed consent before any assessment is performed

Exclusion Criteria:

* Detected M204I/V, N236T, A181V/T mutation in patient serum HBV DNA at Screening visit
* Patient has a history of or clinical signs/symptoms of hepatic decompensation
* Patient has a history of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate the percentage of patients achieving HBV DNA< 300copies/mL at Week 104 in Group I is superior than that in Group II | Week 104

SECONDARY OUTCOMES:
Percentage of patients achieving HBV DNA <60IU/mL (300copies/mL) at Week 52 | week 52
Serum HBV DNA reduction from baseline at week 104 | week 104
Percentage of patients with HBeAg loss & HBeAg seroconversion at week104 in patients with HBeAg positive at baseline | week 104
Percentage of patients with HBV DNA<300copies/mL AND HBeAg loss or seroconversion at Week 104 in patients with positive HBeAg at baseline | week 104
Serum HBV DNA reduction from baseline at week 52 | week 52

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (24):
- China (24):
  - 302 Military Hospital of China, Beijing, Beijing Municipality
  - Beijing Ditan Hospita, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Attached to the Capital Medical University, Beijing, Beijing Municipality
  - BeiJing YouAn Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Department of infectious disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People'S Hospital Under Beijnig University, Beijing, Beijing Municipality
  - The Second Affiliated of ChongQing University of Medical Science, Chongqing, Chongqing Municipality
  - Department of infectious disease, Nanfang Hospital, Guangzhou, Guangdong
  - No. 8 People's Hospital In GuangZhou, Guangzhou, Guangdong
  - The Third Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - No.81 Hospital of PLA, Nanjing, Jiangsu
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shenyang, Liaoning
  - JiNan Infectious Diseases Hospital, Jinan, Shandong
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - No.85 Hospital of PLA, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, XiAn, Shanxi
  - West China Hospital.SiChuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of College of Medicine ，Zhejiang University, Hangzhou, Zhejiang
  - The Sixth People's Hospital of Hangzhou, Hangzhou, Zhejiang

REFERENCES:
- [Background] Keeffe EB, Zeuzem S, Koff RS, Dieterich DT, Esteban-Mur R, Gane EJ, Jacobson IM, Lim SG, Naoumov N, Marcellin P, Piratvisuth T, Zoulim F. Report of an international workshop: Roadmap for management of patients receiving oral therapy for chronic hepatitis B. Clin Gastroenterol Hepatol. 2007 Aug;5(8):890-7. doi: 10.1016/j.cgh.2007.05.004. Epub 2007 Jul 13. PMID 17632041
- [Derived] Huang Q, Zhou B, Cai D, Zong Y, Wu Y, Liu S, Mercier A, Guo H, Hou J, Colonno R, Sun J. Rapid Turnover of Hepatitis B Virus Covalently Closed Circular DNA Indicated by Monitoring Emergence and Reversion of Signature-Mutation in Treated Chronic Hepatitis B Patients. Hepatology. 2021 Jan;73(1):41-52. doi: 10.1002/hep.31240. Epub 2020 Dec 1. PMID 32189364